CLINICAL TRIAL: NCT06456489
Title: Revealing the Potential of Intravenous Pulse Steroid Therapy; Impressive Results in Attaining Remission or Low Disease Activity in Refractory Rheumatoid Arthritis
Brief Title: Pulse Steroid Injection in Refractory Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Prof., Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Al-Azhar University
Record Dates: First submitted 2024-06-01; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Active Rheumatoid Arthritis
MeSH Terms: interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulse steroid solumedrol (Experimental): 125 mg of methylprednisolone IV pulse will be administered for two consecutive days followed by oral steroid for 2 weeks with gradual withdrawal.
  Interventions: Drug: Solumedrol
- without pulse (Placebo Comparator): patients will not receive any additional treatment
  Interventions: Drug: Solumedrol

INTERVENTIONS:
Drug: Solumedrol — 125 mg methylprednisolone intravenous pulse on 2 consecutive days

SUMMARY:
Remission or low disease activity in active rheumatoid arthritis

DETAILED DESCRIPTION:
Assessment of rheumatoid arthritis activity by Disease activity score DAS28, DAS28 Erythrocyte sedimentation rate (ESR), American college of rheumatology (ACR) 20, ACR 50, ACR 70 will be done at baseline and every month for 3 consecutive months for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Refractory rheumatoid arthritis patients

Exclusion Criteria:

* Other connective tissue diseases
* Endocrine diseases such as DM and thyroid disorders

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
remission or low disease activity | 4 months
  Outcome measurements for both groups will be done at baseline and every month for 3 months. DAS28, DAS28 ESR ACR20 ACR50 ACR70

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar Univrsity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided